CLINICAL TRIAL: NCT01409486
Title: Screening for Early Detection and Prevention of Pompe Disease in Israel Using Tandem Mass Spectrometry
Acronym: LC-MS-MS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Hanna Mandel, Rambam Health Care Campus
Other Study IDs: 0290-09-RMB-CTIL
Record Dates: First submitted 2011-07-07; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Pompe Disease
Keywords: Pompe disease; Alpha glucosidase; Newborn screening; Tandem Mass Spectrometry (LC-MS-MS); The study aims:; To establish the control mean values of alpha glucosidase activity in Dry blood spots of Newborn babies from Israel.; To include the alpha glucosidase assay in the newborn screening program in Israel
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Drawing blood spots from Newborns — Dry blood spots would be taken for determination of Alpha Glucosidase activity using LC-MS-MS

SUMMARY:
The aim of the study is:

to develop a comprehensive biochemical assay for detection of Pompe disease (glycogen storage disease type II), to be implemented in the Newborn screening program among the Israeli population.

ELIGIBILITY:
Inclusion Criteria:

* New born babies born during the study period

Exclusion Criteria:

* Premature babies

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 10000 full-term newborns born in Northern Israel
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Identification of the normal mean control value of Alpha glucosidase activity in Dry blood spots among Newborns in Israel | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel